CLINICAL TRIAL: NCT00815061
Title: Epidemiology of Ulcerative Colitis and Crohn's Disease in Non Jewish Israel Population
Status: Withdrawn | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Yaron Niv, Director Department of Gastroenterology, Rabin Medical Center
Other Study IDs: RMC085095CTIL
Record Dates: First submitted 2008-12-24; First posted 2008-12-29 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Ulcerative Colitis; Crohn's Disease
Keywords: prevalence; Incidence; crohn's disease; ulcerative colitis; Epidemiology
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the present study was to describe the incidence and prevalence of IBD in non Jewish Israel population

DETAILED DESCRIPTION:
We are interest to collect the detail of gender, age, duration of the disease and therapy

To obtain the information we wont to contact each physician by e-mail, phone , and fax .

ELIGIBILITY:
Inclusion Criteria:

* ulcertive colitis and crohn's disease patients

Exclusion Criteria:

* N/A

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Crohn's and ulcerative colitis patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Prevalence and incidence of IBD | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Niv, M.D., Principal Investigator — RMC
Locations (1):
- RMC, Petah Tikva, Israel